CLINICAL TRIAL: NCT06011746
Title: Efficacy of Adding Ketamine to Levobupivacaine in Paravertebral Block on Acute and Chronic Pain in Thoracotomy: a Randomized Controlled Double-blinded Trial
Brief Title: Adding Ketamine to Levobupivacaine in Paravertebral Block in Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine Faculty of Medicine Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR244/6/23
Record Dates: First submitted 2023-07-13; First posted 2023-08-25 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Ketamine; Levobupivacaine; Paravertebral Block; Acute Pain; Chronic Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Ketamine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Experimental): patients will receive paravertebral block (19 mL of 0.5% levobupivacaine + 1 ml ketamine (50 mg)).
  Interventions: Drug: Ketamine + Levobupivacaine
- Control Group (Active Comparator): patients will receive paravertebral block (19 mL of 0.5% levobupivacaine + 1 ml normal saline)
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Ketamine + Levobupivacaine — Skin infiltration will be done using 3 ml lidocaine 2% and a 22-gauage block needle will be advanced using the in-plane approach craniocaudally. Once the costotransverse ligament is reached, negative aspiration of blood and air will be confirmed. Under ultrasound visualization, 19 mL of 0.5% levobupivacaine with 1ml ketamine (50mg)
  Arms: Ketamine Group
Drug: Levobupivacaine — Skin infiltration will be done using 3 ml lidocaine 2% and a 22-gauage block needle will be advanced using the in-plane approach craniocaudally. Once the costotransverse ligament is reached, negative aspiration of blood and air will be confirmed. Under ultrasound visualization, 19 mL of 0.5% levobupivacaine with (50mg) or normal saline
  Arms: Control Group

SUMMARY:
To evaluate the role of adding ketamine to levobupivacaine in PVB on acute and chronic pain in thoracotomy

DETAILED DESCRIPTION:
Several adjuvants have been added to them to enhance the effects of those blocks. Dexamethasone, morphine, dexmedetomidine, clonidine, ketamine, and magnesium sulphate are some of them. results are variable.

Ketamine blocks N-Methyl-D-Aspartate (NMDA) receptors in the spinal cord. It is also considered to influence voltage sensitive Calcium ions channels, opioid receptors, and monoaminergic receptors. Therefore, it is considered overall to affect nociception.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Both sexes.
* ASA (American Society of Anesthesiology) physical status II-III.
* Scheduled for open thoracotomy.

Exclusion Criteria:

* Contraindications to or failed paravertebral block .
* Body mass index (BMI) >35 kg/m2.
* The likelihood of postoperative mechanical ventilation.
* Patients with coagulopathy, poorly controlled diabetes mellitus, depression or other psychiatric disorders that required antidepressant drugs, alcohol, or recreational drug addiction.
* Hypersensitivity to ketamine or levobupivacaine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Time to first analgesia | 24 hour postoperatively
  The time till the first rescue of analgesia of morphine. Patients can receive incremental doses of morphine 3 mg intravenously as rescue analgesia if the numeric rating scale (NRS) pain score is > 3.

SECONDARY OUTCOMES:
Total amount of morphine consumption | 24 hour postoperatively
  The total morphine consumption in the 1st 24h postoperative will be recorded. Patients can receive incremental doses of meperidine 0.5 mg/kg intravenously as rescue analgesia if the numeric rating scale (NRS) pain score is > 3.
Pain intensity during rest | 48 hour postoperatively
  Postoperative pain using numeric rating scale at rest and during coughing or movement will be measured at Post-anesthesia care unit, 1h, 2h. 4hr, 6h, 8h, 12h, 18h, 24h, 36h and 48h postoperative.
Pain intensity during deep breathing | 48 hour postoperatively
  Postoperative pain using numeric rating scale at rest and during coughing or movement will be measured at Post-anesthesia care unit, 1h, 2h. 4hr, 6h, 8h, 12h, 18h, 24h, 36h and 48h postoperative.
Incidence of chronic pain | three months postoperatively
  The neuropathic PTPS cases were screened using the grading system for neuropathic pain (GSNP). Positive cases of PTPS with a neuropathic component were grade 2 (probable) or 3 (definite), that is, GSNP ≥2

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author